CLINICAL TRIAL: NCT04296331
Title: Enhancing a Universal Testing and Treatment Strategy in Jail to Promote Viral Load Suppression Among Justice-involved People Living With HIV
Brief Title: HIV Jail POC-AgAB Testings
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Emory University (Other); Unity Health Care, Inc. (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Matthew Akiyama, Assistant Professor of Medicine, Montefiore Medical Center
Other Study IDs: 2020-12451
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: HIV/AIDS
Keywords: Correctional settings; HIV/AIDS; point-of-care testing; rapid Universal Testing and Treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- POC only: Participants who enter the DC Department of Corrections within the first 2 months of the study will be offered opt-out Point-of-Care (POC) rapid testing
  Interventions: Diagnostic Test: POC
- POC + Ag/Ab: Participants who enter the DC Department of Corrections within the third and fourth months of the study will be offered opt-out POC and 4th generation laboratory-based antigen/antibody testing (Ag/Ab)
  Interventions: Diagnostic Test: POC + Ag/Ab
- Ag/Ab only: Participants who enter the DC Department of Corrections within the fifth and sixth months of the study will be offered Ag/Ab testing.
  Interventions: Diagnostic Test: Ag/Ab

INTERVENTIONS:
Diagnostic Test: POC — DC DOC's current testing practice offers opt-out POC testing with the INSTI® finger stick test at entry
  Other Names: INSTI® rapid test
  Groups: POC only
Diagnostic Test: Ag/Ab — The DC DOC will transition from offering their current POC testing upon entry to offering opt-out HIV testing with Ag/Ab: ARCHITECT® laboratory-based test.
  Other Names: Ag/Ab: ARCHITECT® laboratory-based test
  Groups: Ag/Ab only
Diagnostic Test: POC + Ag/Ab — As the DC DOC transitions to utilizing the Ag/Ab: ARCHITECT® laboratory-based test from their current POC testing, jail nurses will offer new entrants op-out testing with the two methods
  Other Names: INSTI® rapid test and ARCHITECT® laboratory-based test
  Groups: POC + Ag/Ab

SUMMARY:
"Enhancing a universal testing and treatment strategy in jail to promote viral load suppression among justice-involved people living with HIV" is an observational research study led by Dr. Matthew Akiyama, MSc of Albert Einstein College of Medicine and Montefiore Medical Center and Dr. Anne Spaulding, MPH of Emory University's Rollins School of Public Health. Due to the high rates of undiagnosed Human Immunodeficiency Virus (HIV) in the correctional setting and the short length of stay in jails, this study aims to evaluate whether care coordination within the D.C. Central Detention Facility (DC DOC) and upon release, including testing procedures and antiretroviral therapy (ART) initiation, can improve the connection of adults (age 18 and over) living with HIV to care in the community.

The researchers will retrospectively look at the aggregate-level de-identified data of roughly 3,000 individuals admitted to the DC DOC over a 6-month period to determine the most effective HIV diagnostic test for routine opt-out testing in the correctional setting. Over the course of these 6 months, the correctional facility will transition from using POC only to POC + antigen/antibody (Ag/Ab), to solely using Ag/Ab, each for a 2-month duration. Individuals from this time period who are identified by corrections staff as HIV-positive either through testing upon admission, their electronic medical record (EMR) or self-report, and have a known release date will be considered eligible for the follow-up study to assess if care coordination is effective in linking others with HIV leaving the DC DOC to care. This follow-up will enroll 100 of these individuals who have consented to participate following their release from the DC DOC, and will consist of a chart review of their DC DOC EMRs and those from their community healthcare provider for up to two years after their release.

DETAILED DESCRIPTION:
This study will be the first to assess the feasibility, process measures, and estimate cost-effectiveness of a rapid Universal Testing and Treatment (rUTT) intervention in a large urban jail located in Washington, DC - 1 of the 50 communities targeted for End the HIV Epidemic (EtHE) efforts. The aim is to determine the most effective HIV diagnostic test to use for routine opt-out testing in the correctional setting.

The investigators hypothesize that the combination of opt-out POC and Ag/Ab tests offered at intake will maximize the yield of PLWH detected, provision of test results, ART initiation, viral suppression, and cost-effectiveness.

The investigators will examine administrative, de-identified, aggregate data for approximately 3000 individuals (based on 500 individuals currently accepting HIV testing per month) over 6 months. For individuals who provide consent to release their jail medical records after incarceration, the investigators will retrieve the mean time from: 1) positive test to receipt of test results, 2) receipt of test results to first dose of ART in jail, 3) receipt of post-test counseling to meeting the discharge planner, and 4) ART initiation to viral suppression defined as a viral load <200 copies/mL. The investigators will calculate the implementation costs of each strategy using observation of staff time, market values for items used in the intervention, and process measure data collected through chart review (for individuals who consent to release their jail medical records after incarceration). Units of resource items, such as staff time and diagnostic tests, will be multiplied by their unit costs to calculate total costs.

This protocol does not constitute research involving prisoners (as outlined by the U.S. Department of Health & Human Services Office for Human Research Protections - https://www.hhs.gov/ohrp/regulations-and-policy/guidance/faq/prisoner-research/index.html) since the investigators will not be:

1. Obtaining identifiable private data or information about prisoner subjects through intervention or interaction with them while incarcerated.
2. Seeking the informed consent of prisoners to be subjects in research;
3. Using, studying or analyzing, for research purposes, identifiable private information about prisoners, or identifiable specimens obtained from prisoners; or
4. Surveying prisoners for this research study.

The overarching goal of this pilot study is to assess 3 HIV testing strategies as the entry point into a rUTT jail-based intervention to promote HIV viral suppression among individuals with undiagnosed and diagnosed HIV infections. Among individuals within the DC Department of Corrections (DC DOC) the investigators will examine whether opt-out Point-of-Care (POC) rapid testing, 4th generation laboratory-based antigen/antibody testing (Ag/Ab), or POC and Ag/Ab testing are most effective in identifying HIV infection upon entry into the jails, linking persons to care and obtaining viral load suppression. During the medical intake, jail nurses will sequentially use, for 2 month each: 1. POC only; 2. POC + Ag/Ab; 3. Ag/Ab only as part of standard clinical care (POC: INSTI® rapid test; Ag/Ab: ARCHITECT® laboratory-based test). Upon anticipation of release, those who are on ART will be invited to participate in a follow-up study regarding their coordination of care while in the DC DOC system and post-release, as well as their current viral load status.

The specific aims are: (1) Compare the feasibility of 3 testing strategies using administrative, de-identified, aggregate data to measure the number/percentage of entrants who do not opt out of testing and receive their test results in jail. (2) Compare 3 testing strategies for time to return of preliminary and confirmed test results, jail-based ART initiation (or reinitiation in known PLWH), and referral to discharge planners among justice-involved PLWH who consent to release their jail medical records after incarceration. (3) Assess the cost of implementing each testing strategy and relative cost-effectiveness of the 3 testing strategies in terms of process measures, time to ART initiation, and viral suppression.

Setting and location The DC DOC is a large urban jail with nearly 8000 intakes per year and an average daily population of approximately 2000 individuals. It is estimated that the HIV prevalence in this system is approximately 4% with a mean of 60 known PLWH in the population at any given time. About 1-3 new HIV diagnoses are made each month with the current POC HIV testing program in place. The patient population is predominantly racial/ethnic minorities (97% overall; 88% Black, 20% Hispanic - not mutually exclusive due to more than 1 race/ethnicity), and 91% are at or below the 200% poverty level (HRSA, 2017). As part of the Unity Health Care (UHC) clinical program, individuals with newly diagnosed HIV will be offered rapid ART initiation, ideally within 24-72 hours of diagnosis with an integrase inhibitor-based regimen as per Department of Health and Human Services(DHHS) guidelines ("Guidelines",2019). Individuals who are known to be HIV-positive through the electronic medical record (EMR) or self-report do not undergo HIV testing. For those who are ART-experienced, the individual's existing ART regimen is restarted. If ART-naïve, an integrase inhibitor-based regimen will be started within 24-72 hours. Community follow-up is offered within 1-2 weeks of reentry and supported by jail discharge planners and community health workers (CHWs). UHC recently began a new 5-year contract to provide jail health services, ensuring a consistent healthcare provider for the duration of this study. DC has expanded Medicaid, which is an essential to developing an rUTT model since it is imperative to ensure no break in ART coverage. Potential participants for this study will be recruited from the DC DOC system

It is estimated that aggregate-level data will be collected for 3,000 individuals who are admitted to the DC DOC system over the 6-month study period and accept HIV testing upon entry. Of those tested, preliminary eligibility will be based on the following criteria:

1. Admitted to DC DOC between October 14th, 2019 and October 31st, 2020
2. Has initiated ART by time of release
3. Being HIV-positive: confirmed either through HIV testing upon entry, was known to be HIV-positive through the EMR, or self-reported being HIV-positive

For the past 12 years DC DOC has offered opt-out POC testing with the INSTI® finger stick test at entry. During booking (in the intake medical evaluation unit, prior to processing individuals into jail) jail nurses will sequentially use, for 2 month each: 1. POC only; 2. POC + Ag/Ab; 3. Ag/Ab only as part of standard clinical care (POC: INSTI® rapid test; Ag/Ab: ARCHITECT® laboratory-based test). To assist UHC with this transition, the investigators have secured in-kind donation of INSTI® rapid test kits (see letter of support). Over 6 months of testing the investigators anticipate approximately 3000 individuals will be tested (based on 500 individuals currently accepting HIV testing per month). The number of new HIV diagnoses that will be made is not known; however, the investigators anticipate the number will be higher using Ag/Ab testing than the 1-3 new diagnoses that are made each month using the current POC rapid testing strategy.

After each of the 3 testing phases the project team will request, from DC DOC, data from their EMR. Specifically, they will request administrative, de-identified, aggregate data that does not contain any of the 18 Health Insurance Portability and Accountability Act (HIPAA) identifiers for: 1) the total number of entrants, 2) the number of entrants with HIV test results (indicating they have not opted out of testing), 3) the number of post-test counseling visits (indicating receipt of test results), 4) the number of positive HIV tests, and 5) the median and mean length of stay for the entire population. The individuals for whom these data are available and are on ART at time of jail release are considered "EMR-eligible participants." Aggregate-level data will be collected on all individuals admitted to DC DOC beginning January 15th, 2019.

Participants for the post-release portion of the study will be recruited at exit from the DC DOC system. Currently the DC DOC provides all patients who are on ART with a 30-day supply upon release. Inmates who are released and have entered the jail during the study period will receive an invitation letter to participate in the study that will be attached to their 30-day supply of ART, which they will pick up at release.

'Invitation to Participate Letters' from UHC will inform EMR-eligible participants that they may be eligible to participate in a paid observational research study about the effectiveness of opt-out rUTT strategies for HIV (see attached letter). Potentially eligible participants are instructed to contact the UHC research coordinator (RC) if they are interested in being a part of the study, or to find out more information. The letter will state that for this observational study participants will only have to continue their standard HIV care with their provider. They will only have to meet with the study team once in order to conduct the eligibility screening and sign the informed consent authorizing the study team to receive the participants EMR from DC DOC and their community provider for two years following their release.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to DC DOC between October 14th, 2019 and October 31st, 2020
* Has initiated ART by time of release
* Being HIV-positive: confirmed either through HIV testing upon entry, was known to be HIV-positive through the EMR, or self-reported being HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals admitted to DC DOC between October 14th, 2019 and October 31st, 2020
Sampling Method: Non-Probability Sample
Enrollment: 6613 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
HIV diagnostic test effectiveness | 6 months
  To determine the most effective HIV diagnostic test for routine opt-out testing in the correctional setting

SECONDARY OUTCOMES:
Linkage to care | 6 months
  Compare 3 testing strategies for time to return of preliminary and confirmed test results, jail-based ART initiation(or reinitiation in known PLWH),and referral to discharge planners among justice-involved PLWH who consent to release their jail medical records after incarceration
Cost-effectiveness | 6 months
  Assess the cost of implementing each testing strategy and relative cost-effectiveness of the 3 testing strategies in terms of process measures, time to ART initiation, and viral suppression

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Akiyama, MD, MSc, Principal Investigator — Montefiore Medical Center
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: What is 'Ending the HIV Epidemic: A Plan for America' — https://www.hiv.gov/federal-response/ending-the-hiv-epidemic/overview
- See also: Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents with HIV. U.S. Department of Health and Human Services website. — https://clinicalinfo.hiv.gov/sites/default/files/guidelines/archive/AdultandAdolescentGL_2021_08_16.pdf